CLINICAL TRIAL: NCT01102478
Title: A Single Dose, 4-Period, 2-Treatment Replicate Design Bioequivalency Study of Losartan Potassium/Hydrochlorothiazide Tablets 100 mg/25 mg Under Fasting Conditions
Brief Title: Bioequivalency Study of Losartan Potassium/Hydrochlorothiazide 100 mg/25 mg Tablet Under Fasted Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Elizabeth Ernst, Roxane Laboratories, Inc.
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LOHY-T100/25-PVFS-1
Record Dates: First submitted 2010-04-09; First posted 2010-04-13 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — hydrochlorothiazide, losartan drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: losartan potassium / hydrochlorothiazide — 100 mg / 25 mg tablet
  Other Names: Hyzaar

SUMMARY:
The objective of this study was to prove the bioequivalence of Losartan Potassium/Hydrochlorothiazide 100/25 mg tablet under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening.

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.
* History of allergic or adverse response to losartan potassium hydrochlorothiazide or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2005-02; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Bioequivalence determined by statistical comparison Cmax | 25 days

CONTACTS AND LOCATIONS:
Overall Officials: Daniel V Freeland, D.O., Principal Investigator — CEDRA Clinical Research, LLC
Locations (1):
- CEDRA Clinical Research, LLC, Austin, Texas, United States